CLINICAL TRIAL: NCT04139226
Title: A Phase 1, Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of CC-11050 After Single and Multiple Doses of CC-11050 and Evaluate CC-11050 Pharmacokinetics Under Fasted and Fed Conditions and After Administration of CC-11050 Alone Compared to Co-administration With a Proton Pump Inhibitor in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability Pharmacokinetics, and Pharmacodynamics of a New Spray Dried Dispersion (SDD) Formulation of CC-11050 After Single Dose of CC-11050 and to Evaluate the Pharmacokinetics of CC-11050 Under Fasted and Fed Conditions and After Coadministration With Omeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-11050-CP-010; U1111-1240-5519 (Other: WHO)
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
Keywords: CC-11050; Safety; Healthy Subjects
MeSH Terms: interventions — CC-11050

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-11050 (Experimental): Part 1: Single Ascending Dose Part 2: drug-drug interaction/ food effect (DDI/FE)
  Interventions: Drug: CC-11050

INTERVENTIONS:
Drug: CC-11050 — CC-11050

SUMMARY:
This is a two-part study to be conducted at single study center, (additional center(s) may be selected if needed) to assess the safety, tolerability, PK and PD parameters for a new SDD formulation of CC-11050 in healthy subjects. The effects of a high-fat meal and omeprazole will also be assessed. Blood samples will be collected at prespecified times for PK, clinical laboratory safety assessments, PD (Part 1 only), and/or exploratory analyses. Safety will be monitored throughout the study from the time the ICF is signed through study completion.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is a male, or a non-pregnant and non-nursing female between 18 and 55 years, inclusive, of age at the time of signing the Informed Consent Form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject has a BMI ≥ 18 and ≤ 33 kg/m2 at screening.
5. Female subject

   1. Must have a negative pregnancy test
   2. If postmenopausal: must have follicular stimulating hormone (FSH) test result >40 IU/L and a negative pregnancy test
6. Contraception Requirements:

   Must comply with the following acceptable forms of contraception. All females of childbearing potential (FCBP) must use one of the approved contraceptive2 options described below while taking CC-11050 and for at least 28 days after administration of the CC-11050 dose. At the time of study entry, and at any time during the study when a FCFP's contraceptive measures or ability to become pregnant changes, the Investigator will educate the subject regarding contraception options and the correct and consistent use of effective contraceptive methods in order to successfully prevent pregnancy. A FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below: Option 1: One highly effective method (eg, hormonal contraception [oral, injection, implant, transdermal patch, vaginal ring]; intrauterine device; tubal ligation; or partner's vasectomy) and 1 additional form (latex condom or any nonlatex condom not made of natural [animal] membrane [eg, polyurethane], diaphragm, sponge).

   OR Option 2: Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane) PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
7. A male subject must:

   a. Practice true abstinence3 (which must be reviewed on a monthly basis and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or female of FCBP while participating in the study, during dose interruptions, and for at least 28 days after the dose of IP, even if he has undergone a successful vasectomy.
8. Subject has clinical laboratory safety test results that are within normal limits (WNL) or acceptable to the Investigator.
9. Subject is afebrile (febrile is defined as ≥ 38°C or ≥100.4°F), with supine systolic blood pressure ≥ 90 and ≤ 150 mm Hg, supine diastolic blood pressure ≥ 50 and ≤ 90 mm Hg, and pulse rate ≥ 40 and ≤ 100 beats per minute at screening
10. Subject is in good health as determined by past medical history, PE, vital signs, 12-lead ECG, and clinical laboratory safety tests. Clinical laboratory safety tests (ie, hematology, chemistry, and urinalysis) and 12-lead ECGs must be WNL or clinically acceptable as judged by the Investigator.
11. Subject has a normal or clinically acceptable 12-lead ECG at screening. In addition:

    * If male, the subject has a QTcF value ≤ 450 msec at screening
    * If female, the subject has a QTcF value ≤ 470 msec at screening

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject is pregnant or breastfeeding.
5. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever was longer).
6. Subject has used moderate or strong CYP3A4/5 inducers and/or inhibitors (including St. John's wort) within 30 days prior to dosing. The Indiana University P450 Drug Interactions Flockhart Table™ may be consulted for a list of such medications.
7. Subject has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure. A subject with an appendectomy and/or cholecystectomy may be included.
8. Subject has donated blood or plasma within 8 weeks before dose administration to a blood bank or blood donation center.
9. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dose administration, or positive drug screening test reflecting consumption of illicit drugs unless positive drug screen is due to prescription drug use that is approved by the Investigator and the Medical Monitor.
10. Subject has a history of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 1 year before dose administration, or a positive alcohol screen.
11. Subjects smokes more than 10 cigarettes per day, or the equivalent in order tobacco products (self-reported).
12. Subject has had a positive result to the test for human immunodeficiency virus (HIV) antibodies at Screening.

    • Chronic or resolved Hepatitis B or Hepatitis C are acceptable only if sequelae are limited to hepatic involvement and its consequent comorbidities. (ie, vasculitis, clinically significant globulinemia, etc. are unacceptable).
13. Subject has received a live vaccination (excluding seasonal flu vaccination) within 30 days of dosing.
14. Used prescribed systemic or topic medication within 30 days of the first dose administration
15. Used any non-prescribed systemic or topic medication (including vitamin/mineral supplements, and herbal medicines, eg, St. John's Wort) within 14 days of the first dose administration, unless Sponsor agreement is obtained.
16. History of significant multiple and/or severe allergies (e.g., food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or.
17. Subject is, for any reason, deemed by the Investigator to be inappropriate for this study, including a subject who is unable to communicate or to cooperate with the investigator or the clinical staff.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values (as specified by the criteria in Section 10.3), regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax | Up to approximately 8 days at hour 192
  Maximum plasma concentration of drug
Pharmacokinetics - Tmax | Up to approximately 8 days at hour 192
  Time to reach maximum observed plasma concentration
Pharmacokinetics - AUC 0-∞ | Up to approximately 8 days at hour 192
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacokinetics - AUC 0-t | Up to approximately 8 days at hour 192
  Area under the plasma concentration-time curve from time zero to the last measured time point
Pharmacokinetics - AUC 0-24 | Up to approximately 8 days at hour 192
  Area under the plasma concentration-time curve from time zero to 24 hours
Pharmacokinetics - AUC 0-12 | Up to approximately 8 days at hour 192
  Area under the plasma concentration-time curve from time zero to 12 hours
Pharmacokinetics - t1/2 | Up to approximately 8 days at hour 192
  Terminal elimination half-life
Pharmacokinetics - Accumulation index (Rac) | Up to approximately 8 days at hour 192
  Accumulation ratio
Pharmacokinetics - CL/F | Up to approximately 8 days at hour 192
  Apparent total plasma clearance when dosed orally
Pharmacokinetics - Vz/F | Up to approximately 8 days at hour 192
  Apparent volume of distribution when dosed orally

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States